CLINICAL TRIAL: NCT06126835
Title: Ozanimod Pregnancy Safety Study in Pregnant Women With Ulcerative Colitis and Their Offspring
Brief Title: A Study to Evaluate the Safety of Ozanimod Exposure During Pregnancy in Women With Ulcerative Colitis and Their Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-025
Record Dates: First submitted 2023-10-06; First posted 2023-11-13 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ozanimod exposed
  Interventions: Drug: Ozanimod
- Conventional therapy exposed
  Interventions: Drug: Conventional therapy
- Advanced therapy exposed
  Interventions: Drug: Advanced therapy

INTERVENTIONS:
Drug: Ozanimod — Women with UC exposed to ozanimod during pregnancy
  Groups: Ozanimod exposed
Drug: Conventional therapy — Women with UC exposed to conventional therapy (aminosalicylates, azathioprine, or mercaptopurine) during pregnancy
  Groups: Conventional therapy exposed
Drug: Advanced therapy — Women with UC exposed to advanced therapy (infliximab, adalimumab, golimumab, vedolizumab, ustekinumab, tofacitinib, cyclosporine, or tacrolimus) during pregnancy
  Groups: Advanced therapy exposed

SUMMARY:
The purpose of this retrospective observational cohort study is to assess pregnancy and infant outcomes in three groups: the first is women with ulcerative colitis (UC) who were exposed to ozanimod during pregnancy; the second is women with UC exposed to conventional therapy during pregnancy; the third is women with UC exposed to advanced therapy during pregnancy. This study will use data from a large US healthcare claims database.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 49 years on date of conception
* Date of conception between June 1, 2021 and September 1, 2030
* Continuous medical and pharmacy coverage for a minimum of 6 months prior to date of last menstrual period through the end of the pregnancy episode
* Diagnosis of UC during the 12 months prior to conception through the end of the first trimester

Exclusion Criteria:

* • Pregnancies exposed to any known teratogens and the exposure falls within the period of 5 half-lives prior to the estimated date of conception through the end of the first trimester (assessed via the presence of national drug codes or medical procedure codes)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult women with UC who became pregnant between June 1, 2021 and September 1, 2030
Sampling Method: Non-Probability Sample
Enrollment: 2828 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2031-05-31 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of major congenital malformations among infants | Up to 10 years
  To estimate and compare the prevalence of major congenital malformations among infants born to pregnant women with UC who were exposed to ozanimod during first trimester relative to the prevalence among (i) infants born to women with UC exposed to conventional UC treatments and (ii) infants born to women with UC exposed to advanced UC treatment during first trimester of pregnancy.

SECONDARY OUTCOMES:
Number of spontaneous abortions | Up to 10 years
Number of stillbirths | Up to 10 years
Number of participants with pre-eclampsia | Up to 10 years
Number of participants with eclampsia | Up to 10 years
Number of preterm births | Up to 10 years
Number of infants small for gestational age | Up to 10 years
Number of serious or opportunistic infections in liveborn infants up to 1 year of age | Up to 10 years
Number of infant postnatal growth deficiencies | Up to 10 years
Number of infant developmental deficiencies | Up to 10 years
Number of neonatal hospitalizations | Up to 10 years
Number of infant deaths | Up to 10 years
Number of neonatal deaths | Up to 10 years
Number of perinatal deaths | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- OptumInsight Life Sciences Inc, Eden Prairie, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts